CLINICAL TRIAL: NCT01245127
Title: Ilaris (Canakinumab) in the Schnitzler Syndrome. A Case Series.
Brief Title: Ilaris (Canakinumab) in the Schnitzler Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S52762
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2010-11

CONDITIONS: Schnitzler Syndrome
Keywords: Schnitzler syndrome
MeSH Terms: conditions — Schnitzler Syndrome | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canakinumab (Experimental): * Canakinumab 150 mg (or 2 mg/kg for patients weighing <40kg) every 8 weeks over a 6 months treatment period (i.e., weeks 0, 8, 16 and 24).
  * At Day 7, patients who show an improvement, but not a clinical remission, will be given another 150 mg (or 2 mg/kg for patients weighing <40 kg) injection and continue at 300 mg (or 4 mg/kg for patients weighing <40 kg) every 8 weeks beginning at Week 8.
  * Patients who show no improvement of symptoms and signs of Schnitzler's syndrome will not receive any additional canakinumab dose and will be offered corticosteroid therapy. These patients will return for a follow-up visit 2 weeks later (Day 21) for safety reasons and will be discontinued from the trial.
  * If a patient flares twice during the study, physician may optionally change the dosing frequency to every 4 weeks.
  Interventions: Drug: Ilaris

INTERVENTIONS:
Drug: Ilaris — * Canakinumab 150 mg (or 2 mg/kg for patients weighing <40kg) every 8 weeks over a 6 months treatment period (i.e., weeks 0, 8, 16 and 24).
  * At Day 7, patients who show an improvement, but not a clinical remission, will be given another 150 mg (or 2 mg/kg for patients weighing <40 kg) injection and continue at 300 mg (or 4 mg/kg for patients weighing <40 kg) every 8 weeks beginning at Week 8.
  * Patients who show no improvement of symptoms and signs of Schnitzler's syndrome will not receive any additional canakinumab dose and will be offered corticosteroid therapy. These patients will return for a follow-up visit 2 weeks later (Day 21) for safety reasons and will be discontinued from the trial.
  * If a patient flares twice during the study, physician may optionally change the dosing frequency to every 4 weeks.

SUMMARY:
Schnitzler syndrome:

Schnitzler syndrome is a rare disabling autoinflammatory syndrome characterized by a chronic urticarial rash and monoclonal gammopathy, accompanied by intermittent fever, arthralgia or arthritis or bone pain. Diagnostic criteria have been established. The disease never remits spontaneously. Although there is no standard of care, there have been promising developments in therapeutic options, especially anti-interleukin-1 therapy. Anakinra, a synthetic analogue of the endogenous interleukin-1 receptor antagonist, has caused rapid clinical remission in 24 patients with Schnitzler syndrome. However, to sustain remission, continuous daily administration (100 mg sc) is required. The level of monoclonal protein does not decrease. Side effects of anakinra include painful injection site reactions and neutropenia.

Interleukin-1 and the autoinflammatory diseases:

As a key proinflammatory cytokine mediating local and systemic responses to infection and tissue injury, interleukin-1 can induce a range of responses, including fever, pain sensitization, bone and cartilage destruction, and the acute-phase inflammatory response. The so-called autoinflammatory diseases are mediated entirely by interleukin-1; reducing interleukin-1 activity brings about a rapid and sustained remission. Autoinflammatory diseases include relatively uncommon disorders such as familial Mediterranean fever, adult and juvenile Still's disease, the hyper-IG D syndrome, Behçet's syndrome, the cryoporin-associated periodic syndrome (CAPS), deficiency of the interleukin-1 receptor antagonist (DIRA) and Schnitzler's syndrome. Some common conditions such as gout and type 2 diabetes, are also likely to be autoinflammatory diseases.

Canakinumab:

Canakinumab (Ilaris, Novartis Pharma) is a fully human anti-interleukin-1-bèta monoclonal antibody. Treatment with subcutaneous canakinumab (150 mg) once every 8 weeks was associated with a rapid remission of symptoms in the great majority of children and adults with CAPS. Serum inflammatory markers quickly returned to normal. In general, the side effects seen in this small study (35 patients) were not serious, though suspected infections ware significantly more prevalent in patients receiving canakinumab than in those receiving placebo. The prolonged duration of action of canakinumab and low incidence of injection-site reactions may confer certain advantages over other interleukin-1 inhibitors (anakinra and rilonacept), since both are frequently associated with injection-site reactions, and both require more frequent administration (daily for anakinra and weekly for rilonacept).

Canakinumab was approved for the treatment of CAPS by the US Food and Drug Administration in June 2009 and by the European Medicines Agency in October 2009.

Canakinumab is currently being evaluated for its potential in the treatment of systemic-onset juvenile idiopathic arthritis, diabetes mellitus, and difficult-to-treat gouty arthritis.

DETAILED DESCRIPTION:
Description of the study:

Objectives:

* Primary objective: To evaluate if canakinumab 150mg every 8 weeks can induce and maintain clinical remission in patients with the Schnitzler syndrome.
* Secondary objectives:

  * To test if canakinumab 150mg can induce a complete clinical response at Day 7.
  * To assess if addition canakinumab 150mg given at Day 7 for patients demonstrating only a partial response can induce a complete clinical response at Day 14.
  * To evaluate if canakinumab 300mg every 8 weeks can maintain clinical remission in those patients who required canakinumab 150 mg additional dose on Day 7 and achieved clinical remission at Day 14.
  * To evaluate the safety of canakinumab treatment in patients with the Schnitzler syndrome.
  * To assess the changes in C-reactive protein (CRP) levels during the treatment period.

Study rationale:

Although no standard therapy has been established for the Schnitzler syndrome, given the rarity of this auto-inflammatory syndrome, reports on the use of Anakinra, a synthetic analog of the endogenous interleukin-1 receptor antagonist, have been encouraging. However, side effects (including local infusion site reactions and neutropenia) and the need for daily sc administration have hampered its use. The anti-interleukin-1-inhibitor canakinumab may constitute an effective and more convenient alternative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Schnitzler syndrome after withdrawal of anakinra or tapering of corticosteroids.
* Male and female patients at least 18 years of age at the time of screening visit.
* Signed patient informed consent
* Negative QuantiFERON test or negative Purified Protein Derivative (PPD) test (<5 mm induration) at screening or within 1 month prior to the screening visit, according to Belgium guidelines. Patients with a positive PPD test (=5 mm induration) at screeninig may be enrolled only if they have a negative chest x-ray or negative QuantiFERON test (QFT-TB G In-Tube).
* Adequate contraception in females of childbearing potential.

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot)
* Serologic evidence of active hepatitis B or C infection
* Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose.
* History of significant medical conditions, which in the investigator's opinion would exclude the patient from participating in this trial.
* History of recurrent and/or evidence of active bacterial, fungal or viral infection(s).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: body temperature, arthralgia, urticaria, fatigue, C-reactive protein | 28 weeks
  Primary parameters include body temperature, arthralgia, urticaria, fatigue, C-reactive protein.
  Response is defined as:
  1. Resolution of periodic fever: no body temperatures above 38.2°C
  2. Resolution of chronic urticaria
  3. Normalization of CRP
  4. Resolution of chronic arthralgia/arthritis and bone pains.

SECONDARY OUTCOMES:
Tolerability: injection site reactions | 28 weeks
  tolerability, including injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vanderschueren, MD, PhD, Principal Investigator — General Internal Medicine, UZ Gasthuisberg, Leuven
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] de Koning HD, Bodar EJ, van der Meer JW, Simon A; Schnitzler Syndrome Study Group. Schnitzler syndrome: beyond the case reports: review and follow-up of 94 patients with an emphasis on prognosis and treatment. Semin Arthritis Rheum. 2007 Dec;37(3):137-48. doi: 10.1016/j.semarthrit.2007.04.001. Epub 2007 Jun 21. PMID 17586002
- [Background] Besada E, Nossent H. Dramatic response to IL1-RA treatment in longstanding multidrug resistant Schnitzler's syndrome: a case report and literature review. Clin Rheumatol. 2010 May;29(5):567-71. doi: 10.1007/s10067-010-1375-9. Epub 2010 Feb 1. PMID 20119842
- [Background] Dybowski F, Sepp N, Bergerhausen HJ, Braun J. Successful use of anakinra to treat refractory Schnitzler's syndrome. Clin Exp Rheumatol. 2008 Mar-Apr;26(2):354-7. PMID 18565263
- [Background] Gilson M, Abad S, Larroche C, Dhote R. Treatment of Schnitzler's syndrome with anakinra. Clin Exp Rheumatol. 2007 Nov-Dec;25(6):931. No abstract available. PMID 18173934
- [Background] Frischmeyer-Guerrerio PA, Rachamalla R, Saini SS. Remission of Schnitzler syndrome after treatment with anakinra. Ann Allergy Asthma Immunol. 2008 Jun;100(6):617-9. doi: 10.1016/S1081-1206(10)60064-6. No abstract available. PMID 18592830
- [Background] Lachmann HJ, Kone-Paut I, Kuemmerle-Deschner JB, Leslie KS, Hachulla E, Quartier P, Gitton X, Widmer A, Patel N, Hawkins PN; Canakinumab in CAPS Study Group. Use of canakinumab in the cryopyrin-associated periodic syndrome. N Engl J Med. 2009 Jun 4;360(23):2416-25. doi: 10.1056/NEJMoa0810787. PMID 19494217
- [Derived] Vanderschueren S, Knockaert D. Canakinumab in Schnitzler syndrome. Semin Arthritis Rheum. 2013 Feb;42(4):413-6. doi: 10.1016/j.semarthrit.2012.06.003. Epub 2012 Aug 15. PMID 22901459